CLINICAL TRIAL: NCT02607423
Title: Role of Early 18F-FDG-PET/CT Scan in Predicting Mediastinal Downstaging With Neoadjuvant Chemotherapy in Resectable Stage III A NSCLC
Brief Title: Fludeoxyglucose F-18 PET/CT in Predicting Response to Chemotherapy in Patients With Stage IIIA Non-small Cell Lung Cancer That Can Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study failed to meet its accrual targets.
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA5123; NCI-2015-01054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5123 (Other: ECOG-ACRIN Cancer Research Group); EA5123 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stage IIIA Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Fluorodeoxyglucose F18; Gemcitabine; Pemetrexed; Magnetic Resonance Spectroscopy

ARMS (1):
- Diagnostic (18F-FDG PET/CT) (Experimental): Patients undergo fludeoxyglucose F-18 PET/CT at baseline and after course 1 of chemotherapy. Patients undergo 1 of 3 chemotherapy regimens at the discretion of the investigator.
  CHEMOTHERAPY REGIMEN 1: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, and 8. Patients also receive cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  CHEMOTHERAPY REGIMEN 2: Patients receive docetaxel IV over 60 minutes and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  CHEMOTHERAPY REGIMEN 3: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Radiation: Fludeoxyglucose F-18; Drug: Gemcitabine Hydrochloride; Drug: Pemetrexed Disodium; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo 18F-FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Radiation: Fludeoxyglucose F-18 — Undergo 18F-FDG PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Procedure: Positron Emission Tomography — Undergo 18F-FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) works in predicting response to chemotherapy in patients with stage IIIA non-small cell lung cancer that can be removed by surgery (resectable). Performing diagnostic procedures, such as fludeoxyglucose F-18 PET/CT, after one course of chemotherapy may help doctors predict a patient's response to treatment earlier and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether percent change in maximum standardized uptake value (SUVmax) on FDG-PET/CT from T0 to T1 measured on mediastinal lymph nodes can predict mediastinal downstaging in patients with stage IIIA-N2 non-small cell lung cancer (NSCLC) treated with neoadjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the predictive accuracy for mediastinal downstaging of two other FDG-PET/CT-based markers measured on mediastinal lymph nodes: SUVmax at T1 and change of SUVmax from T0 to T1.

II. To evaluate the predictive accuracy for mediastinal downstaging of the FDG-PET/CT-based markers measured on the primary tumor, include percent change of peak standardized uptake value (SUVpeak) (based on PET Response Criteria in Solid Tumors [PERCIST] criteria), total lesion glycolysis (TLG) and metabolic tumor volume (MTV) from T0 to T1.

III. To evaluate whether percent change in SUVmax on FDG-PET/CT from T0 to T1 measured on mediastinal lymph nodes can predict overall survival (OS).

OUTLINE:

Patients undergo fludeoxyglucose F-18 PET/CT at baseline and after course 1 of chemotherapy. Patients undergo 1 of 3 chemotherapy regimens at the discretion of the investigator.

CHEMOTHERAPY REGIMEN 1: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, and 8. Patients also receive cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

CHEMOTHERAPY REGIMEN 2: Patients receive docetaxel IV over 60 minutes and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

CHEMOTHERAPY REGIMEN 3: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have stage IIIA non-small cell lung cancer (T1-3N2) per American Joint Committee on Cancer (AJCC) 7th edition and must be considered to be surgically resectable
* Patients must be assessed by surgeons and are considered surgically resectable
* Mediastinal nodal metastases (N2) disease must be confirmed histologically
* Easter Cooperative Oncology Group (ECOG) performance status 0 or 1
* Required imaging studies obtained within four weeks prior to registration
* White blood cell (WBC) >= 4000 mm^3 or granulocyte count at least 2,000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 10.0g/dL
* Total bilirubin < 1.5 mg/dL
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) < 3 x upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3 x ULN
* Alkaline phosphatase < 3 x ULN
* Calculated/estimated or measured creatinine clearance at least 50 ml/min; note: creatinine clearance should be calculated using the Cockcroft-Gault formula; patients who will receive pemetrexed/cisplatin therapy must be obtained within 2 weeks of registration
* Patients cannot have hormonal cancer therapy or radiation therapy as prior cancer treatment within 5 years of registration; (prior surgery, biologic therapy, hormonal therapy, or radiation therapy for a malignancy over 5 years prior to enrollment that is not considered cured is acceptable)
* Patients must not have any history of other cancer within 5 years from registration with the exception of in situ carcinoma of the cervix, in situ carcinoma of the breast or completely resected non-melanoma skin cancer
* Patients may not have received prior chemotherapy or radiation therapy for lung cancer
* Patients with a history of myocardial infarction are eligible if the event occurred > 6 months prior to entry
* Patients must not have any clinically significant ongoing, active or serious infection, symptomatic or uncontrolled congestive heart failure, active angina, symptomatic or uncontrolled cardiac arrhythmia or any other medical condition or psychiatric illness/social situations that would limit compliance with study requirements
* Patents must have no contraindication to cisplatin chemotherapy including no clinically significant hearing loss unless willing to accept the potential of further loss of hearing, no symptomatic peripheral neuropathy
* Women must not be pregnant or breast-feeding
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study
* Patients must not have received any study therapies prior to registration
* Pemetrexed/cisplatin therapy; note: patients who will receive pemetrexed/cisplatin therapy must meet all eligibility criteria below:

  * Patients assigned to pemetrexed/cisplatin therapy must NOT have squamous cell histology
  * Calculated creatinine clearance must be obtained within 2 weeks of registration and calculated creatinine clearance (CrCl) must be >= 45mL/min using the standard Cockcroft and Gault formula, or the measured glomerular filtration rate (GFR) using the appropriate radiolabeled method (51-CrEDTA or Tc99m-DTPA) must be used to calculate CrCl
* Patients should have no contraindications for FDG-PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-19 (Estimated); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of mediastinal downstaging | Up to 9 weeks
  The predictive accuracy of the percent change in SUVmax on FDG-PET/CT from T0 to T1 measured on mediastinal lymph nodes will be estimated by the area under a receiver operating characteristic (ROC) curve (AUC) with a 95% confidence interval (CI). The AUC will be estimated empirically. The reference standard for the ROC analysis will be the presence or absence of mediastinal downstaging, as assessed by thoracotomy, mediastinoscopy, mediastinotomy, endoscopic bronchoscopic ultrasound (EBUS), or endoscopic ultrasound (EUS).

SECONDARY OUTCOMES:
Change of SUVmax | Baseline to 3 weeks
  The predictive accuracy of the change in SUVmax on FDG-PET/CT from T0 to T1 measured on mediastinal lymph nodes will be estimated by the ROC AUC with a 95% CI. The AUC will be estimated empirically.
Overall survival | Up to 5 years
  Time-dependent ROC analysis will be used to determine the predictive accuracy of percent change in SUVmax on FDG-PET/CT from T0 to T1 measured on mediastinal to predict overall survival.
Percent change of metabolic tumor volume | Baseline to 3 weeks
  The predictive accuracy of percent change of metabolic tumor volume from T0 to T1 from primary tumor will be measured by the ROC AUC with a 95% CI. The AUC will be estimated empirically.
Percent change of SUVpeak | Baseline to 3 weeks
  The predictive accuracy of percent change of SUVpeak from T0 to T1 from primary tumor will be measured by the ROC AUC with a 95% CI. The AUC will be estimated empirically.
Percent change of TLG | Baseline to 3 weeks
  The predictive accuracy of percent change of TLG from T0 to T1 from primary tumor will be measured by the ROC AUC with a 95% CI. The AUC will be estimated empirically.
SUVmax | At 3 weeks
  The predictive accuracy of SUVmax at T1 will be estimated by the ROC AUC with a 95% CI. The AUC will be estimated empirically.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States